CLINICAL TRIAL: NCT00462384
Title: An Open-label, Multi-center Study to Demonstrate Correction of Anemia and to Assess the Maintenance of Hemoglobin Levels Using Subcutaneous Once Monthly Injections of Mircera in Pre-dialysis Patients With Chronic Kidney Disease
Brief Title: A Study of Subcutaneous Mircera for the Treatment of Anemia in Pre-Dialysis Participants With Chronic Kidney Disease.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision unrelated to safety or efficacy
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20659
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Methoxy Polyethylene Glycol-epoetin Beta (Experimental): Methoxy polyethylene glycol-epoetin beta will be administered subcutaneously every 4 weeks (at Weeks 4, 8, 12, 16, 20, 24, 28 and 32). The starting dose will be 1.2 micrograms per kilogram (mcg/kg) body weight. Thereafter, throughout the duration of study the dose adjustments will be performed depending on the hemoglobin value.
  Interventions: Drug: Methoxy Polyethylene Glycol-epoetin Beta

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-epoetin Beta — Methoxy polyethylene glycol-epoetin beta will be administered subcutaneously every 4 weeks (at Weeks 4, 8, 12, 16, 20, 24, 28 and 32). The starting dose will be 1.2 mcg/kg body weight. Thereafter, throughout the duration of study the dose adjustments will be performed depending on the hemoglobin value.
  Other Names: Mircera; RO0503821

SUMMARY:
This single arm study will assess the efficacy and safety of subcutaneous Mircera for correction of anemia in participants with chronic kidney disease who are not on dialysis and are not treated with erythropoiesis-stimulating agents (ESA). Eligible participants will receive Mircera by monthly subcutaneous injections, dependent on body weight (with a starting dose of 1.2 micrograms/kilogram [mcg/kg]). The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease, stage 3 or 4;
* anemia (baseline hemoglobin between 9 and 11 grams per deciliter [g/dL]).

Exclusion Criteria:

* previous therapy with ESA within 12 weeks prior to screening;
* significant acute or chronic bleeding such as overt gastrointestinal bleeding;
* red blood cell transfusions within 8 weeks before screening;
* active malignant disease (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (8):
  - HUS
  - Joensuu
  - Jyväskylä
  - Kajaani
  - Kotka
  - Porvoo
  - Tampere
  - Turku
- Latvia (5):
  - Jūrmala
  - Liepāja
  - Riga
  - Valmiera
  - Ventspils
- Norway (5):
  - Hønefoss
  - Lillehammer
  - Oslo
  - Stavanger
  - Trondheim

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta: Methoxy polyethylene glycol-epoetin beta was administered subcutaneously every 4 weeks (at Weeks 4, 8, 12, 16, 20, 24, 28 and 32). The starting dose was 1.2 micrograms per kilogram (mcg/kg) body weight. Thereafter, throughout the duration of study the dose adjustments were performed depending on the hemoglobin value.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Started | 39
Completed | 30
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: Safety population: included all participants who were treated with at least one dose of the study medication.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta: Methoxy polyethylene glycol-epoetin beta was administered subcutaneously every 4 weeks (at Weeks 4, 8, 12, 16, 20, 24, 28 and 32). The starting dose was 1.2 mcg/kg body weight. Thereafter, throughout the duration of study the dose adjustments were performed depending on the hemoglobin value.
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (18.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Concentration Between Baseline and the Efficacy Evaluation Period (EEP)
Description: The baseline hemoglobin was defined as the mean of the assessments recorded during the screening period (Weeks -2 and 0). EEP was the first 8 weeks (Weeks 29 to 36) following the 28 weeks dose titration period. EEP hemoglobin was defined as the mean of the assessments recorded during the EEP.
Time Frame: Baseline (Week -2 to 0) and EEP (Weeks 29 to 36)
Population: Intent to treat (ITT) population: included all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta and for whom data for at least one study variable was available.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 39
grams per deciliter (g/dL) | 1.32 (0.88)

2. Secondary Outcome: Time to Achievement of Response
Description: Time to achievement of response was the time (number of days) required to achieve hemoglobin levels within the range of 11.0 to 13.0 g/dL.
Time Frame: Baseline to Week 40
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 39
days | 24.6 (20.53)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentration Within Hemoglobin Range 11.0 to 13.0 g/dL Throughout the EEP
Description: EEP was the first 8 weeks (Weeks 29 to 36) following the 28 weeks dose titration period. The percentage of participants whose hemoglobin concentrations remained within the range of 11.0-13.0 g/dL at all assessments throughout the EEP is presented.
Time Frame: EEP (Weeks 29 to 36)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 39
percentage of participants | 53.9

4. Secondary Outcome: Percentage of Participants Maintaining Average Hemoglobin Concentration Within Hemoglobin Range 11.0 to 13.0 g/dL During the EEP
Description: EEP was the first 8 weeks (Weeks 29 to 36) following the 28 weeks dose titration period. The percentage of participants whose average hemoglobin concentration was within the range of 11.0-13.0 g/dL during the EEP is presented.
Time Frame: EEP (Weeks 29 to 36)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 39
percentage of participants | 66.7

5. Secondary Outcome: Time Spent in Hemoglobin Range of 11.0 to 13.0 g/dL During the EEP
Description: EEP was the first 8 weeks (Weeks 29 to 36) following the 28 weeks dose titration period.
Time Frame: EEP (Weeks 29 to 36)
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 39
days | 42.5 (13.96)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 40
Description: Safety population
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Serious Adverse Events (participants affected / at risk) | 11/39
Other Adverse Events (participants affected / at risk) | 11/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=39)
Angina pectoris (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bronchitis (Infections and infestations) | 1
Otitis media chronic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1
Azotaemia (Renal and urinary disorders) | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Foot amputation (Surgical and medical procedures) | 1
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=39)
Urinary tract infection (Infections and infestations) | 4
Insomnia (Psychiatric disorders) | 2
Urine odour abnormal (Renal and urinary disorders) | 2
Hypertension (Vascular disorders) | 5

LIMITATIONS AND CAVEATS:
This study was terminated early due to strategic decision unrelated to safety or efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.